CLINICAL TRIAL: NCT05646719
Title: Randomized, Double-Masked, Placebo-Controlled, Multicenter, Phase 3 Study of the Safety and Efficacy of Nyxol (Phentolamine Ophthalmic Solution 0.75%) as a Single Agent and With Adjunctive Low-Dose Pilocarpine Hydrochloride Ophthalmic Solution 0.4% in Subjects With Presbyopia
Brief Title: Safety and Efficacy of Nyxol Eye Drops as a Single Agent and With Adjunctive Low-Dose Pilocarpine Eye Drops in Subjects With Presbyopia
Acronym: VEGA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXP-301 (VEGA-2)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-07

CONDITIONS: Presbyopia
Keywords: Nyxol; Presbyopia; Pilocarpine
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Nyxol + low dose pilocarpine (Experimental): Nyxol (phentolamine ophthalmic solution) 0.75% Pilocarpine (0.4%)
  Interventions: Drug: Phentolamine Opthalmic Solution 0.75%; Drug: Low dose pilocarpine
- Nyxol + low dose pilocarpine vehicle (Experimental): Nyxol (phentolamine ophthalmic solution) 0.75% Pilocarpine vehicle
  Interventions: Drug: Phentolamine Opthalmic Solution 0.75%; Other: Low dose pilocarpine vehicle
- Placebo + low dose pilocarpine (Experimental): Placebo Pilocarpine (0.4%)
  Interventions: Other: Placebo; Drug: Low dose pilocarpine
- Placebo + low dose pilocarpine vehicle (Experimental): Placebo Pilocarpine vehicle
  Interventions: Other: Placebo; Other: Low dose pilocarpine vehicle
- Nyxol (Experimental): Nyxol (phentolamine ophthalmic solution) 0.75%
  Interventions: Drug: Phentolamine Opthalmic Solution 0.75%
- Nyxol placebo (Experimental): Nyxol placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phentolamine Opthalmic Solution 0.75% — phentolamine ophthalmic solution 0.75% (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol
  Arms: Nyxol; Nyxol + low dose pilocarpine; Nyxol + low dose pilocarpine vehicle
Other: Placebo — Vehicle for Phentolamine Ophthalmic Solution
  Other Names: Phentolamine Ophthalmic Solution Vehicle
  Arms: Nyxol placebo; Placebo + low dose pilocarpine; Placebo + low dose pilocarpine vehicle
Drug: Low dose pilocarpine — Pilocarpine hydrochloride ophthalmic solution 0.4%
  Other Names: Pilocarpine; LDP
  Arms: Nyxol + low dose pilocarpine; Placebo + low dose pilocarpine
Other: Low dose pilocarpine vehicle — Vehicle for low dose pilocarpine
  Arms: Nyxol + low dose pilocarpine vehicle; Placebo + low dose pilocarpine vehicle

SUMMARY:
The objectives of this study are:

To evaluate the safety and efficacy of Nyxol alone and with adjunctive low dose pilocarpine to improve distance-corrected near visual acuity (DCNVA) in subjects with presbyopia.

DETAILED DESCRIPTION:
This is a Randomized, Double-Masked, Placebo-Controlled, Multicenter, Phase 3 Study of the Safety and Efficacy of Nyxol (Phentolamine Ophthalmic Solution 0.75%) as a Single Agent and With Adjunctive Low-Dose Pilocarpine Hydrochloride Ophthalmic Solution 0.4% in Subjects With Presbyopia

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 40 and ≤ 64 years of age.
2. BCDVA of 0.1 LogMAR (20/25 Snellen equivalent) or better in each eye in photopic conditions.
3. DCNVA of 0.4 LogMAR (20/50 Snellen equivalent) or worse but not > 0.7 LogMAR (20/100 Snellen equivalent) in photopic conditions in each eye and binocularly.
4. For subjects who depend on reading glasses or bifocals, binocular best-corrected near VA is 0.1 LogMAR (20/25 Snellen equivalent) or better.
5. Photopic PD of ≥ 3 mm in either eye.

Exclusion Criteria:

Ophthalmic (in either eye):

1. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind within 7 days of Screening until study completion, with the exception of lid scrubs with OTC products and artificial tears as specified in Exclusion # 2 below.
2. Use of any OTC artificial tears (preserved or unpreserved) during Visit days or 15 min before or after instillation of study medication.
3. Current use of any topical ophthalmic therapy for dry eye.
4. Tear break-up time of < 5 seconds or corneal fluorescein staining Grade ≥ 2 in the inferior zone or Grade ≥ 1 in the central zone using the National Eye Institute scale..
5. Clinically significant ocular disease that might interfere with the study as deemed by the Investigator.
6. Recent or current evidence of ocular infection or inflammation in either eye.
7. Any history of herpes simplex or herpes zoster keratitis.
8. Known allergy, hypersensitivity, or contraindication to any component of the phentolamine, pilocarpine, or vehicle formulations.
9. Prior participation in a study involving the use of Nyxol for the treatment of presbyopia.
10. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal.
11. Ocular trauma within 6 months prior to Screening.
12. Ocular surgery or any ocular laser treatment within 6 months prior to Screening.
13. Subjects with surgical monovision, multifocal or extended depth of focus intraocular lenses (IOLs) are excluded.
14. History of any traumatic (surgical or nonsurgical) or nontraumatic condition affecting the pupil or iris.
15. Contact lens wear on the day of any study visit and contact lenses must be removed for home dosing and for at least 10 minutes following dosing.

    Systemic:
16. Known hypersensitivity or contraindication to alpha- and/or beta-adrenoceptor antagonists .
17. Known hypersensitivity or contraindication to any systemic cholinergic parasympathomimetic agent.
18. Clinically significant systemic disease that might interfere with the study as deemed by the judgment of the Investigator.
19. Initiation of treatment with, or any changes to, the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to Screening or during the study.
20. Participation in any investigational study within 30 days prior to Screening.
21. Females of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.
22. Resting HR outside the range of 50 to 110 beats per min.
23. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Phoenix, AZ, Phoenix, Arizona
  - Azusa, CA, Azusa, California
  - Newport Beach, CA, Newport Beach, California
  - Northridge, CA, Northridge, California
  - Delray Beach, FL, Delray Beach, Florida
  - Longwood, FL, Longwood, Florida
  - Roswell, GA, Roswell, Georgia
  - Lake Villa, IL, Lake Villa, Illinois
  - Pittsburg, KS, Pittsburg, Kansas
  - Shawnee Mission, KS, Shawnee Mission, Kansas
  - Bloomington, MN, Bloomington, Minnesota
  - Chesterfield, MO, Chesterfield, Missouri
  - Kansas City, MO, Kansas City, Missouri
  - Saint Louis, MO, St Louis, Missouri
  - Rochester, NY, Rochester, New York
  - Smithtown, NY, Smithtown, New York
  - Garner, NC, Garner, North Carolina
  - Fargo, ND, Fargo, North Dakota
  - Athens, OH, Athens, Ohio
  - Cranberry Township, PA, Cranberry Township, Pennsylvania
  - New Freedom, PA, New Freedom, Pennsylvania
  - Sioux Falls, SD, Sioux Falls, South Dakota
  - Memphis, TN, Memphis, Tennessee
  - Austin, TX, Austin, Texas
  - Houston, TX, Houston, Texas
  - San Antonio, TX, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nyxol + Low Dose Pilocarpine | Nyxol + Low Dose Pilocarpine Vehicle | Placebo + Low Dose Pilocarpine | Placebo + Low Dose Pilocarpine Vehicle
Started | 83 | 84 | 83 | 83
Completed | 78 | 80 | 79 | 82
Not Completed | 5 | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Nyxol + Low Dose Pilocarpine | Nyxol + Low Dose Pilocarpine Vehicle | Placebo + Low Dose Pilocarpine | Placebo + Low Dose Pilocarpine Vehicle | Total
Number analyzed (Participants) | 82 | 81 | 82 | 82 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Modified intent to treat population used
  years | 54.2 (5.22) | 55.4 (5.15) | 54.3 (5.92) | 54.4 (4.99) | 54.6 (5.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 64 | 61 | 236
  Male | 26 | 26 | 18 | 21 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 12 | 18 | 56
  Not Hispanic or Latino | 67 | 70 | 70 | 64 | 271
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 1 | 1 | 0 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 16 | 15 | 10 | 57
  White | 64 | 64 | 65 | 69 | 262
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 82 | 82 | 327

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With ≥ 15 Letters of Improvement in Photopic Binocular DCNVA and With < 5 Letters of Loss in Photopic Binocular BCDVA in Nyxol-treated Subjects
Description: The primary efficacy endpoint is the percent of subjects with ≥ 15 letters of improvement in photopic binocular DCNVA and with < 5 letters of loss in photopic binocular BCDVA from Baseline at 30 min post-LDP/vehicle comparing subjects treated with Nyxol + LDP to subjects treated with placebo + LDP vehicle at Visit 5 (Stage 2 Day 8).
Time Frame: Baseline at 30 min post-LDP/vehicle comparing subjects treated with Nyxol + LDP to subjects treated with placebo + LDP vehicle at Visit 5 (Stage 2 Day 8)
Population: Modified Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Nyxol + Low Dose Pilocarpine | Nyxol + Low Dose Pilocarpine Vehicle | Placebo + Low Dose Pilocarpine | Placebo + Low Dose Pilocarpine Vehicle
Number analyzed (Participants) | 78 | 80 | 79 | 82
Participants | 27 | 31 | 16 | 22
Statistical Analysis 1: Comparison: Nyxol + Low Dose Pilocarpine vs Placebo + Low Dose Pilocarpine Vehicle; Test type: Superiority; p < 0.01, t-test, 2 sided; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.23 to 4.20]
Statistical Analysis 2: Comparison: Nyxol + Low Dose Pilocarpine vs Placebo + Low Dose Pilocarpine Vehicle; Test type: Superiority; Odds Ratio (OR) = 1.44

ADVERSE EVENTS:
Time Frame: Through study completion; approximately 43 days.
Description: Study used clinicaltrials.gov definitions
Arm/Group | Nyxol + Low Dose Pilocarpine | Nyxol + Low Dose Pilocarpine Vehicle | Placebo + Low Dose Pilocarpine | Placebo + Low Dose Pilocarpine Vehicle
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80 | 0/81 | 0/82
Other Adverse Events (participants affected / at risk) | 13/79 | 12/80 | 18/81 | 13/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nyxol + Low Dose Pilocarpine (N=79) | Nyxol + Low Dose Pilocarpine Vehicle (N=80) | Placebo + Low Dose Pilocarpine (N=81) | Placebo + Low Dose Pilocarpine Vehicle (N=82)
Instillation site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Instillation site foreign body sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Instillation site irritation (General disorders) | 9 (9) | 9 (9) | 13 (13) | 11 (11)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05646719/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05646719/SAP_001.pdf